CLINICAL TRIAL: NCT01487473
Title: The Effects of Mindfulness-Based Stress Reduction on Attention and Pain-related Symptoms in Chronic Pain Patients: A Randomized Controlled Trial
Brief Title: The Effects of Mindfulness-Based Stress Reduction on Attention and Pain-related Symptoms in Chronic Pain Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: York University (Other)
Collaborators: Mount Sinai Hospital, Canada (Other); Wasser Pain Management Centre (Unknown); Rasch Foundation (Unknown)
Responsible Party: Principal Investigator, Nicholas Cepeda, Associate Professor, York University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: FWA00003852
Record Dates: First submitted 2011-12-05; First posted 2011-12-07 (Estimated); Last update posted 2014-02-13 (Estimated); Status verified 2014-02

CONDITIONS: Pain
Keywords: Meditation; Mindfulness; Attention; Chronic Pain; Depression; Anxiety; Stress; Acceptance; Pain intensity; Pain disability
MeSH Terms: conditions — Pain; Chronic Pain; Depression; Anxiety Disorders | interventions — Mindfulness-Based Stress Reduction

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Mindfulness-Based Stress Reduction (Active Comparator)
  Interventions: Behavioral: Mindfulness-Based Stress Reduction
- Waitlist Control (No Intervention)

INTERVENTIONS:
Behavioral: Mindfulness-Based Stress Reduction — An 8-week structured group program that was developed to improve psychological and physical symptoms associated with pain. It incorporates a variety of mindfulness meditation exercises including mindful yoga, sitting meditation, and body scan to facilitate attention, acceptance, and awareness of one's experiences.
  Other Names: MBSR
  Arms: Mindfulness-Based Stress Reduction

SUMMARY:
The main purpose of this study is to determine the degree to which Mindfulness-Based Stress Reduction, a group-based psychological therapy that includes mindfulness meditation exercises, reduces depression, anxiety, stress, pain intensity, and interference of pain with daily life among adult chronic pain patients.

The second purpose is to examine the role of attention in improving psychological and physical health for chronic pain patients.

ELIGIBILITY:
Inclusion Criteria:

* Adult chronic pain patients who are proficient in English
* Capable of interacting with others in a group setting
* Capable of working with a computer

Exclusion Criteria:

* Alcohol or drug abuse (past history is acceptable as long as their situation has been stable for at least 3 months)
* Psychiatric psychosis (patients who have a past history of schizophrenia are eligible as long as they are currently stable)
* Current major depressive disorder
* Current severe social phobia
* At immediate risk for suicide
* Cerebral lesions or tumors (unless medically and cognitively stable)
* Neurological disease
* Medically unstable
* Cognitively unstable
* Previously participated in a mindfulness meditation program

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2011-12; Primary Completion 2013-11 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
Pain disability and Attention | Baseline, immediately following treatment, and at 3 months follow up
  Change in pain disability assessed by the Pain Disability Index (PDI).
  Change in attention assessed by an adapted version of the Change Blindness Task

SECONDARY OUTCOMES:
Depression | Baseline, immediately following treatment, and at 3 months follow up
  Change in depression assessed by the Depression, Anxiety, and Stress Scale 21 (DASS-21)
Anxiety | Baseline, immediately following treatment, and at 3 months follow up
  Change in anxiety assessed by the Depression, Anxiety, and Stress Scale 21 (DASS-21)
Stress | Baseline, immediately following treatment, and at 3 months follow up
  Change in stress assessed by the Depression, Anxiety, and Stress Scale 21 (DASS-21)
Mindfulness | Baseline, immediately following treatment, and at 3 months follow up
  Change in mindfulness assessed by the Five Facet Mindfulness Questionnaire (FFMQ) and Mindful Attention Awareness Scale (MAAS)
Acceptance | Baseline, immediately following treatment, and at 3 months follow up
  Change in acceptance assessed by the Chronic Pain Acceptance Questionnaire (CPAQ)
Pain Intensity | Baseline, immediately following treatment, and at 3 months follow up
  Change in pain intensity assessed by the Short-form McGill Pain Questionnaire (SF-MPQ-2).

CONTACTS AND LOCATIONS:
Overall Officials: Nicholas Cepeda, PhD, Principal Investigator — York University; Allan Gordon, MD, Principal Investigator — MOUNT SINAI HOSPITAL; Denise Paneduro, PhD student, Study Director — York University
Locations (1):
- Mount Sinai Hospital, Toronto, Ontario, Canada